CLINICAL TRIAL: NCT06965361
Title: Stromal Tumor-Infiltrating Lymphocyte Levels Are Associated With Immune Checkpoint Proteins In Triple Negative Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Acronym: TIL; PD1; PDL1
Status: Completed | Type: Observational
Sponsor: Ziauddin University (Other)
Collaborators: Jinnah Sindh Medical University (Other)
Responsible Party: Principal Investigator, Shamim Mushtaq, Professor, Ziauddin University
Other Study IDs: 1730120SMBIO; 20-11952/NRPU/RGM/R&D/HEC (Other Grant/Funding Number: Higher Education Commission)
Record Dates: First submitted 2025-04-23; First posted 2025-05-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: carboplatin-based NACT regimen; tumor-infiltrating lymphocytes; Programmed cell death-1; Programmed cell death Ligand-1; lymphocyte activation gene-3; Triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Doxorubicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- A+T group and A+T+C group: All TNBC patients included in the study received at least four cycles of NACT regimens and were classified into two groups: anthracycline-containing, taxane- (A+T group) and anthracycline/taxane/carboplatin (A+T+C group) combinations
  Interventions: Drug: carboplatin; Device: carboplatin

INTERVENTIONS:
Drug: carboplatin — carboplatin use due to its effectiveness in increasing pathological complete remission (pCR) rates and improving survival outcomes
  Other Names: Doxorubicin
Device: carboplatin — used in the treatment of triple-negative breast cancer (TNBC) due to its effectiveness in achieving pathological complete response (pCR) and breast-conserving surgery (BCS) rates.
  Other Names: Carpsol®

SUMMARY:
The goal of this observational study is to learn about the effects of neoadjuvant chemotherapy (NACT) anthracycline-containing, taxane- (Intervention A +T) and anthracycline/taxane /carboplatin (Intervention A+T+C) treatment in young (age; 24-45 years) Triple Negative Breast Cancer (TNBC) female Patients by evaluating Stromal tumor-infiltrating lymphocytes (TILs) Programmed cell death-1 (PD-1), its ligand (PD-L1) and lymphocyte activation gene-3 (LAG-3) checkpoint proteins within tumor.

The main question it aims to answer is:

Does TILs are the most reliable immune markers and are significantly associated with PD-1, PD-L1 and LAG-3 in carboplatin based NACT treated (Intervention A+T+C) group of TNBC patients? Participants (TNBC Patients) already taking intervention A+T and A+T+C as part of their regular medical care for TNBC.

DETAILED DESCRIPTION:
Stromal tumor-infiltrating lymphocytes (TILs) are currently being considered as a prognostic factor in triple-negative breast cancer (TNBC) and their association with the tumor immune microenvironment is less clear. To address this knowledge gap, investigators aimed to evaluate the expression and association of Programmed cell death-1 (PD-1), its ligand (PD-L1) and lymphocyte activation gene-3 (LAG-3) checkpoint proteins with TILs in neoadjuvant chemotherapy (NACT) treated TNBC patients.

Patients (n=54; aged;24-45 years) were classified into two groups: thirty-nine received anthracycline-containing, taxane- (A+T group) and fifteen received anthracycline/taxane /carboplatin (A+T+C group) in combinations. Immunohistochemistry (IHC) staining was used for the evaluation of PD-1, PD-L1 and LAG-3. However, TIL assessment was done by hematoxylin and eosin (H&E)-staining in TNBC patient's biopsies who received NACT.

ELIGIBILITY:
Inclusion Criteria:

* Female (aged 24-45 years) TNBC patients
* Diagnosed TNBC Patients with immunohistochemistry (IHC) negative test for estrogen receptor (ER), progesterone receptor (PR), and HER-2
* Patients with and without metastases

Exclusion Criteria:

* Patients who had a history of other malignant tumors
* Patients who did not complete NAC.

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with diagnosed TNBC (Age;24-45 years)
Study Population: Karachi subset of population
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Stromal tumor-infiltrating lymphocyte levels are associated with immune checkpoint proteins in triple negative breast cancer patients receiving neoadjuvant chemotherapy | From enrollment to the end of treatment received at least four cycles of NACT regimens. One cycle last for 21 days.
  The TILs levels were evaluated on Hematoxylin-eosin-stained (H&E) tissue sections as percentages and three predefined categories were used: Low TIL scores of 0-10%, intermediate 11-40% and high TIL > 40%.

SECONDARY OUTCOMES:
Evaluation of PD-1, PD-L1 and LAG-3 in triple negative breast cancer patients receiving neoadjuvant chemotherapy | From enrollment to the end of treatment received at least four cycles of NACT regimens. One cycle last for 21 days.
  Patients (n=54; aged;24-45 years) were classified into two groups: thirty-nine received anthracycline-containing, taxane- (A+T group) and fifteen received anthracycline/taxane /carboplatin (A+T+C group) in combinations. Immunohistochemistry (IHC) staining was used for the evaluation of PD-1, PD-L1 and LAG-3. However, TIL assessment was done by hematoxylin and eosin (H&E)-staining in TNBC patient's biopsies who received NACT.

CONTACTS AND LOCATIONS:
Overall Officials: Shamim Mushtaq, PhD, Principal Investigator — Ziauddin University
Locations (1):
- Shamim, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loibl S, Weber KE, Timms KM, Elkin EP, Hahnen E, Fasching PA, Lederer B, Denkert C, Schneeweiss A, Braun S, Salat CT, Rezai M, Blohmer JU, Zahm DM, Jackisch C, Gerber B, Klare P, Kummel S, Schem C, Paepke S, Schmutzler R, Rhiem K, Penn S, Reid J, Nekljudova V, Hartman AR, von Minckwitz G, Untch M. Survival analysis of carboplatin added to an anthracycline/taxane-based neoadjuvant chemotherapy and HRD score as predictor of response-final results from GeparSixto. Ann Oncol. 2018 Dec 1;29(12):2341-2347. doi: 10.1093/annonc/mdy460. PMID 30335131
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC6369970/